CLINICAL TRIAL: NCT05996744
Title: A Phase 2/3 Single-Arm, Open-label Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Obeldesivir in Pediatric Participants With COVID-19
Brief Title: Study of Obeldesivir in Children and Adolescents With COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated by Sponsor; the decision was not due to any safety findings.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-611-6464; 2023-503282-27 (Other: European Medicines Agency)
Record Dates: First submitted 2023-08-14; First posted 2023-08-18 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg (Experimental): Participants received ODV tablets (350 mg twice daily) for 5 days.
  Interventions: Drug: Obeldesivir
- ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg (Experimental): Participants received ODV tablets (175 mg twice daily) for 5 days.
  Interventions: Drug: Obeldesivir

INTERVENTIONS:
Drug: Obeldesivir — Tablet administered orally with or without food
  Other Names: GS-5245

SUMMARY:
The goal of this clinical study is to learn more about the safety and tolerability of obeldesivir (ODV) in children and adolescents with coronavirus disease 2019 (COVID-19).

The primary objectives are to evaluate the plasma pharmacokinetics (PK), safety and tolerability of ODV in pediatric participants with COVID-19.

DETAILED DESCRIPTION:
Pediatric participants will be enrolled as follows:

* Cohort 1: ≥ 6 years to < 18 years and weight ≥ 40 kg
* Cohort 2: ≥ 6 years to < 18 years and weight ≥ 20 kg to < 40 kg
* Cohort 3: ≥ 2 years to < 18 years and weight ≥ 12 kg to < 20 kg
* Cohort 4: ≥ 28 days to < 18 years and weight ≥ 3 kg to < 12 kg
* Cohort 5: ≥ 14 days to < 28 days of age, gestational age (GA) ≥ 37 weeks and weight ≥ 2.5 kg
* Cohort 6: 0 days to < 14 days of age, GA ≥ 37 weeks and birth weight ≥ 2.5 kg
* Cohort 7: 0 days to < 56 days of age, GA < 37 weeks and birth weight ≥ 1.5 kg

ELIGIBILITY:
Key Inclusion Criteria:

* Individual or legal guardian willing and able to provide written informed consent prior to performing study procedures. Individuals will provide assent, if possible, in accordance with local requirements and investigator's discretion.
* Aged < 18 years who meet one of the following weight criteria and gestational age (GA) criteria where applicable:

  * Cohort 1: ≥ 6 years to < 18 years and weight ≥ 40 kg
  * Cohort 2: ≥ 6 years to < 18 years and weight ≥ 20 kg to < 40 kg
  * Cohort 3: ≥ 2 years to < 18 years and weight ≥ 12 kg to < 20 kg
  * Cohort 4: ≥ 28 days to < 18 years and weight ≥ 3 kg to < 12 kg
  * Cohort 5: ≥ 14 days to < 28 days of age, GA ≥ 37 weeks and weight ≥ 2.5 kg
  * Cohort 6: 0 days to < 14 days of age, GA ≥ 37 weeks and birth weight ≥ 2.5 kg
  * Cohort 7: 0 days to < 56 days of age, GA < 37 weeks and birth weight ≥ 1.5 kg
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) or an alternative molecular diagnostic assay ≤ 5 days before screening.
* Initial onset of coronavirus disease 2019 (COVID-19) signs/symptoms ≤ 5 days before screening with ≥ 1 sign/symptom such as fever, cough, fatigue, shortness of breath, sore throat, headache, myalgia/arthralgia present at screening.
* Presence of ≥ 1 characteristic or underlying medical condition associated with an increased risk of developing severe illness due to COVID-19 per protocol.

Key Exclusion Criteria:

* Anticipated access to and use of authorized or approved COVID-19 therapies during the current COVID-19 illness < 5 days after screening (therapies including but not limited to nirmatrelvir/ritonavir, molnupiravir, intravenous remdesivir (RDV), monoclonal antibodies).
* Vaccination for SARS-CoV-2 or self-reported history of SARS-CoV-2 infection < 4 months prior to screening.
* Received any approved, authorized, or investigational direct acting antiviral drug against SARS-CoV-2 for the treatment of COVID-19 < 28 days or < 5 half-lives, whichever is longer, before enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (18):
  - Trinity Clinical Research, LLC, Centreville, Alabama
  - Advanced Research Center, Inc., Anaheim, California
  - Stanford University Medical Center, Palo Alto, California
  - UF Health- Shands Hospital, Gainesville, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - Accel Research Sites Network - Nona Pediatric Center, Orlando, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Santos Research Center, Tampa, Florida
  - Pas Research, Tampa, Florida
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - Pas Research, Las Vegas, Nevada
  - Velocity Clinical Research -Albuquerque, Albuquerque, New Mexico
  - Child Health Care Associates, East Syracuse, New York
  - Velocity Clinical Research, Charleston, Charleston, South Carolina
  - PanAmerican Clinical Research, LLC, Brownsville, Texas
  - Texas Children's Hospital, Houston, Texas
  - The University of Texas Medical School at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT05996744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The study was terminated early after 3 participants were enrolled. The decision to terminate the study early was not due to any safety concerns.
Period: Overall Study
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who enrolled in the study and received the study drug were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Customized [Count of Participants; unit: Participants]
  ≥ 6 years to < 18 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 3.57 (0.991) | 4.36 (NA) — Since only 1 participant was analyzed, Standard Deviation (SD) cannot be calculated. | 3.84 (0.836)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of GS-441524, Metabolite of Obeldesivir (ODV)
Time Frame: Day 3 (5 to 8 hours postdose) and Day 5 (predose and 15 minutes, 30 minutes, 1 hour, and 4 hours postdose)
Population: All participants who enrolled in the study and received the study drug were included. Participants with available data and for whom plasma concentrations of GS-441524 were available were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
ng/mL
  Day 3 (5 to 8 hours postdose) | 1950 (933) | NA (NA) — The plasma concentration was below the limit of quantification.
  Day 5 (predose) | 79.2 (97.3) | NA (NA) — The plasma concentration was below the limit of quantification.
  Day 5 (15 minutes postdose): number analyzed (Participants) | 1 | 1
  Day 5 (15 minutes postdose) | 8.37 (NA) — Since only 1 participant was analyzed, SD cannot be calculated. | 209 (NA) — Since only 1 participant was analyzed, SD cannot be calculated.
  Day 5 (30 minutes postdose): number analyzed (Participants) | 1 | 0
  Day 5 (30 minutes postdose) | 14.5 (NA) — Since only 1 participant was analyzed, SD cannot be calculated. |
  Day 5 (1 hour postdose): number analyzed (Participants) | 1 | 0
  Day 5 (1 hour postdose) | 510 (NA) — Since only 1 participant was analyzed, SD cannot be calculated. |
  Day 5 (4 hours postdose): number analyzed (Participants) | 1 | 0
  Day 5 (4 hours postdose) | 1610 (NA) — Since only 1 participant was analyzed, SD cannot be calculated. |

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (AEs) by Day 35
Description: Treatment-emergent adverse events are defined as 1 or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
percentage of participants | 0 | 0

3. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities by Day 35
Description: Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of last dose of study drug plus 30 days participants who permanently discontinued study drug.
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
percentage of participants | 0 | 0

4. Secondary Outcome: Time to Sustained Alleviation of Targeted Coronavirus Disease 2019 (COVID-19) Symptoms by Day 35
Description: The time to sustained alleviation of targeted COVID-19 symptoms will be calculated as the last date on which the symptom alleviation is assessed by Day 35 minus the first dose date plus 1 day or Day 34, whichever occurs first. Symptom alleviation is defined as follows: all targeted symptoms scored moderate or severe at baseline are scored as mild or none for at least 48 consecutive hours, and all targeted symptoms scored mild or none at baseline are scored as none for at least 48 consecutive hours; the first day of the 48 consecutive hours will be considered the symptom alleviation date. Targeted symptoms include: stuffy or runny nose, sore throat, shortness of breath, cough, low energy or tiredness, muscle or body aches, headache, chills or shivering, feeling hot or feverish, and nausea.
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
Days | 3.4 (0.47) | 2.5 (NA) — Since only 1 participant was analyzed, SD cannot be calculated.

5. Secondary Outcome: Change From Baseline in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Viral Load at Day 5
Description: Nasal swab samples will be used to assess SARS-CoV-2 viral load.
Time Frame: Baseline, Day 5
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
log10 copies/mL | -0.61 (0.868) | NA (NA) — The viral load assay uses two markers, N1 and N2, to amplify two different regions of the SARS-CoV-2 genome. For the participant in Cohort 2 on Day 5, one marker yielded a positive result and the other a negative result, therefore the assay resulted in an error and the result is inconclusive. There was no numerical result derived on Day 5 for the Cohort 2 participant since the result was inconclusive.

6. Secondary Outcome: Percentage of Participants Who Require Supplemental Oxygen Support by Day 35
Description: Supplemental oxygen support included low flow oxygen, high flow oxygen, noninvasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation.
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
percentage of participants | 0 | 0

7. Secondary Outcome: Palatability for Each Formulation as Measured by Questionnaire Responses Assessed by the Study Participants
Description: A questionnaire was administered to participants to assess the palatability of the formulation. Palatability was assessed by questions about how the study drug tasted.
Time Frame: Day 5
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
Participants
  No Taste | 1 | 0
  Neutral Taste (Maybe Good or Maybe Bad) | 1 | 1

8. Secondary Outcome: Acceptability for Each Formulation as Measured by Questionnaire Responses Assessed by the Study Participants
Description: A questionnaire was administered to participants to assess the acceptability of the formulation. Acceptability was assessed by questions about the size of the drug and how easy it was to swallow the study drug.
Time Frame: Day 5
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
Participants
  Super Easy to Swallow | 1 | 0
  Easy to Swallow | 1 | 0
  Hard to Swallow | 0 | 1
  Size: Okay | 2 | 1

9. Secondary Outcome: Percentage of Participants With Concomitant Use of Medications Other Than Remdesivir (RDV) and Obeldesivir (ODV) for Treatment of COVID-19 by Day 35
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
percentage of participants | 0 | 0

10. Secondary Outcome: Percentage of Participants With COVID-19-Related Hospitalization or All-Cause Death by Day 35
Time Frame: First dose date up to Day 35
Population: All participants who enrolled in the study and received the study drug were included.
Measure: Number; unit: percentage of participants
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
Number analyzed (Participants) | 2 | 1
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 35 days
Description: All-cause mortality and adverse events: All participants who enrolled in the study were included.
Arm/Group | Obeldesivir (ODV) 350 mg Twice Daily, Cohort 1: ≥ 6 Years to < 18 Years and Weight ≥ 40 kg | ODV 175 mg Twice Daily, Cohort 2: ≥ 6 Years to < 18 Years and Weight ≥ 20 kg to < 40 kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT05996744/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT05996744/SAP_001.pdf